CLINICAL TRIAL: NCT01716260
Title: Parasitic Clearance and Recurrence Rates Among Patients With Vivax Malaria on Chloroquine and Primaquine Therapy
Brief Title: Safety and Efficacy of Chloroquine and Primaquine for Vivax Malaria in Bhutan
Status: Completed | Type: Observational
Sponsor: Menzies School of Health Research (Other)
Collaborators: Ministry of Health, Bhutan (Other Government)
Responsible Party: Sponsor
Other Study IDs: Bhutan_APMEN_CQ PQ_2013
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2015-04

CONDITIONS: Vivax Malaria
MeSH Terms: conditions — Malaria, Vivax | interventions — Chloroquine; Primaquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chloroquine and Primaquine: Chloroquine (CQ)10mg/kg for day 1, 2 and 5mg/kg for day 3 Primaquine (PQ)0.25mg/kg/day for 14 days
  Interventions: Drug: Chloroquine; Drug: Primaquine

INTERVENTIONS:
Drug: Chloroquine
Drug: Primaquine

SUMMARY:
This research is intended to study the efficacy of chloroquine (CQ) and primaquine (PQ) for Plasmodium vivax (P.vivax) infection, and also to study the recurrence rate among patients with P.vivax malaria on standard doses of CQ and PQ. For this study, PQ will be withheld for 28 days so as to study the efficacy of CQ alone.

This study will assess whether CQ is still effective against P.vivax or whether there are resistant P.vivax strains in Bhutan.

DETAILED DESCRIPTION:
This study aims to assess the efficacy of Chloroquine alone, withholding Primaquine until day 28. Parasitic clearance and recurrence rates will be recorded. Patients whose blood stage of parasites are not cleared with the standard dose of Chloroquine, or any recurrences before day 28, will be treated with second line treatment (ACT).

The patients blood level of Chloroquine (drug concentration) at the time of a recrudescent infection will de determined to assess whether that could be due to resistance, or due to low level of Chloroquine.

Any relapses occurring after day 28 when not receiving Primaquine, or after completion of Primaquine dosage for a total of 14 days (from day 29 to 42), will be treated with repeat doses of the initial treatment. The recurrence rates will be recorded so as to develop the next phase of the study where the two different doses of Primaquine (high dose vs. low dose) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* >12 months of age
* infection with P.vivax parasitaemia monoinfection
* presence of axillary temperature >37.5 degrees or history of fever during the past 24 hours
* ability to swallow oral medication
* ability and willingness to comply with the study protocol for the duration of the study, including 12 months follow up
* informed consent from the patient/parent/guardian in the case of children

Exclusion Criteria:

* Presence of general danger signs in children aged under 5 years or signs of severe malaria according to the definitions of WHO
* Presence of severe malnutrition (defined as a child whose growth standard is below -3 z-score, has symmetrical oedema involving at least the feet or has a mid-upper arm circumference < 110 mm);
* History of haemolysis or severe anaemia
* Acute anaemia <7 mg/dL
* Presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* Regular medication, which may interfere with antimalarial pharmacokinetics
* History of hypersensitivity reactions or contraindications to any of the medicine(s) being tested or used as alternative treatment(s)
* a positive pregnancy test or lactating

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with P.vivax infections will be recruited from 6 sentinel sites and will be recruited for the study after informed consent is received.
  An amendment has been approved to extend the study to 12 sites.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Chloroquine efficacy for P.vivax infections in Bhutan. | 28 days
  The purpose is to study the efficacy of Chloroquine alone by recording recrudescent rates and parasitic clearance in P.vivax patients who are given a standard dose of Chloroquine treatment.

SECONDARY OUTCOMES:
To study the efficacy of Primaquine. | Patients with recurrence after day 28 will be recorded.
  In this study, Primaquine will be administered on day 28, and any relapse will be recorded to study relapse rates over a 12 month period.

OTHER OUTCOMES:
To assess the feasibility of a 12 month follow-up of patients with vivax malaria in Bhutan. | 12 months
To assess the safety of the currently prescribed CQ and PQ regimens in Bhutan. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Vector Diseases Control Program, Geylegphug, Bhutan